CLINICAL TRIAL: NCT01020617
Title: Association Between the Diet, the Composition of Microbiota of the Intestinal Tract, Human Health and Well-being
Brief Title: The Effect of Probiotics on Low-grade Inflammation, Microbiota and Risk Factors for Metabolic Syndrome in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Danish Medical Research Council (Other); Danisco (Industry)
Responsible Party: Professor Kim Fleischer Michaelsen, University of Copenhagen, Department of Human Nutrition
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: D206 ProTeen
Record Dates: First submitted 2009-11-16; First posted 2009-11-25 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2009-11

CONDITIONS: Metabolic Syndrome; Inflammation; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Inflammation; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Ls-33 — 10~10 CFU/day
  Other Names: L. salivarius Ls-33

SUMMARY:
Metabolic syndrome and thereby obesity is associated with low-grade systemic inflammation and it is likely that this is also the case in children (Ley et al., 2005). It has also been shown that the gut microbiota is different in obese individuals compared to normal weight individuals and that the microbiota seems to have a role in fat storage (Backhead et al, 2004).

Intervention study with overweight and normal weight school age children. The children will be randomised to receive selected probiotics or a placebo. Fecal and blood samples will be collected, and anthropometric measurements (weight, height, skin folds) will be recorded before and after the intervention. The dynamic of the microbiota of the GI will be monitored by molecular methods. Markers of intestinal inflammation (calprotectin) and permeability will be analysed. Blood samples will be analysed to evaluate how the intervention influence the systemic polarization of the immune response by means of cytokine analyses. Furthermore, blood pressure, blood lipid profile and early markers of metabolic syndrome will be evaluated. Hypotheses This study will examine if overweight in children is associated with a different intestinal microbiota and if a change in microbiota caused by probiotics can modify inflammation and risk factors for the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 12-15 years
* IsoBMI>30

Exclusion Criteria:

* Chronical diseases
* Chronical medication

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Microbiota diversity | one year
Inflammation, CRP | 2 months
  high sensitive C-reactive protein

SECONDARY OUTCOMES:
Antropometry | one year
Blood pressure | one year
Blood lipids | one year
Fasting insulin | one year
Fasting glucose | one year
C-reactive protein (CRP) | 6 months
Fecal calprotectin | 7 months
Interleukin-6 (Il-6) | one year
Interleukin-10 (IL-10) | one year
Tumor necrosis factor-alpha(TNF-α) | one year
Adiponectin | one year
Leptin | one year
GIP | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kim F Michaelsen, Professor, Principal Investigator — University of Copenhagen, Department of Human Nutrition
Locations (1):
- Copenhagen University, Frederiksberg, Denmark

REFERENCES:
- [Derived] Larsen N, Vogensen FK, Gobel RJ, Michaelsen KF, Forssten SD, Lahtinen SJ, Jakobsen M. Effect of Lactobacillus salivarius Ls-33 on fecal microbiota in obese adolescents. Clin Nutr. 2013 Dec;32(6):935-40. doi: 10.1016/j.clnu.2013.02.007. Epub 2013 Mar 4. PMID 23510724
- [Derived] Giacco R, Lappi J, Costabile G, Kolehmainen M, Schwab U, Landberg R, Uusitupa M, Poutanen K, Pacini G, Rivellese AA, Riccardi G, Mykkanen H. Effects of rye and whole wheat versus refined cereal foods on metabolic risk factors: a randomised controlled two-centre intervention study. Clin Nutr. 2013 Dec;32(6):941-9. doi: 10.1016/j.clnu.2013.01.016. Epub 2013 Feb 6. PMID 23462537
- [Derived] Gobel RJ, Larsen N, Jakobsen M, Molgaard C, Michaelsen KF. Probiotics to adolescents with obesity: effects on inflammation and metabolic syndrome. J Pediatr Gastroenterol Nutr. 2012 Dec;55(6):673-8. doi: 10.1097/MPG.0b013e318263066c. PMID 22695039